CLINICAL TRIAL: NCT04219930
Title: Biochemical Role of Nucleotide Protein -3 That Activate the Interleukin-1B in Epileptic Children
Brief Title: Nucleotide Protein -3 in Epileptic Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham I El-mahdy, Principal Investigator, Assiut University
Other Study IDs: Epilepsy
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Epilepsy in Children
Keywords: Epilepsy; Children; NLRP3; Interleukin B1; Nuclear Factor-Kappa B
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- epileptic children: fifty patient with epilepsy
  Interventions: Diagnostic Test: Expression of nucleotide protein -3
- Healthy controls: thirty healthy control
  Interventions: Diagnostic Test: Expression of nucleotide protein -3

INTERVENTIONS:
Diagnostic Test: Expression of nucleotide protein -3 — Expression of nucleotide protein -3 will be measured in serum by ELISA

SUMMARY:
Epilepsy is one of common serious neurological malfunction, characterized by recurrent unprovoked seizures. It always accompanied with multitude of complications as cognitive, behavioral, and psychiatric disorders.

Experimental studies and clinical evidence obtained in animal models of epilepsy and human brain specimen from various drug-resistant forms of epilepsy show the activation of the innate and adaptive immunity mechanisms and the induction of the associated inflammatory processes in the epileptogenic foci.

DETAILED DESCRIPTION:
Epilepsy affects approximately 1% of the world population. Lifetime prevalence of childhood and adolescence epilepsy (children <18 years) in Upper Egypt was 9.7/1000, with higher prevalence among children <12 years (10.8/1000).

There is a clear cause for epilepsy in only a minority of the cases, while in up to70% of all case of epilepsy in adults and children, no cause can be discovered. Some of the main causes of epilepsy include: Low oxygen during birth, head injuries that occur during birth or from accidents during youth or adulthood, brain tumors, infections such as meningitis or encephalitis, stroke or any other type of damage to the brain.

A role of inflammatory molecules in the generation of seizures had been first investigated when selected anti-inflammatory treatments, in particular, steroids, immuno-globulins, and adrenocorticotropic hormone (ACTH), were shown to control seizures in pediatric epilepsies refractory to conventional anticonvulsive drugs. In addition, specific epileptic disorders have been associated with the presence of neuronal antigen-directed antibodies in plasma or cerebrospinal fluid (CSF).

A nucleotide-binding oligomerization domains (NODs) are cytosolic proteins that include key regulators of apoptosis and pathogen resistance in mammals and plants. A large number of NODs contain leucine-rich repeats (LRRs), hence referred to as NOD-LRR proteins. The NLRP3 gene provides instructions for making a protein called cryopyrin. Cryopyrin is a member of a family of proteins called nucleotide-binding domain and leucine-rich repeat containing (NLR) proteins. NLR family have two common features: the first is a nucleotide-binding oligomerization domain which is bound by ribonucleotide-phosphates (rNTP) and is important for self-oligomerization. The second is a C-terminal leucine-rich repeat, which serves as a ligand-recognition domain for other receptors (e.g. Toll like receptor (TLR)) or microbial ligands, while NLRP3 has been identified in microglial cells.

ELIGIBILITY:
Inclusion Criteria:

* Epileptic children in Assiut university hospital, pediatric department, neurology unit.

Exclusion Criteria:

* Children with other chronic disease such as liver, kidney or heart disease
* patient who have apparent infection

Ages: 2 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Epileptic children
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
The mean difference of nucleotide protein -3 inflammatory marker expression in epileptic children and controls | Baseline
  better understanding the role of inflammation in pathogenesis of epilepsy in children

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He Q, Jiang L, Man S, Wu L, Hu Y, Chen W. Curcumin Reduces Neuronal Loss and Inhibits the NLRP3 Inflammasome Activation in an Epileptic Rat Model. Curr Neurovasc Res. 2018;15(3):186-192. doi: 10.2174/1567202615666180731100224. PMID 30062967
- [Background] Farghaly WM, Abd Elhamed MA, Hassan EM, Soliman WT, Yhia MA, Hamdy NA. Prevalence of childhood and adolescence epilepsy in Upper Egypt (desert areas). Egypt J Neurol Psychiatr Neurosurg. 2018;54(1):34. doi: 10.1186/s41983-018-0032-0. Epub 2018 Nov 9. PMID 30532513
- [Background] Xu D, Miller SD, Koh S. Immune mechanisms in epileptogenesis. Front Cell Neurosci. 2013 Nov 8;7:195. doi: 10.3389/fncel.2013.00195. eCollection 2013. PMID 24265605